CLINICAL TRIAL: NCT02820896
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Intravenous and Subcutaneous RO7105705 Administered in Healthy Volunteers and Patients With Mild-to-Moderate Alzheimer's Disease
Brief Title: A Study of RO7105705 in Healthy Participants and Participants With Mild-to-Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GN39058
Record Dates: First submitted 2016-06-29; First posted 2016-07-01 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Multiple Dose Placebo IV (Placebo Comparator): Healthy participants or participants with Alzheimer's disease will receive multiple doses of matching placebo IV QW, a total of 4 doses.
  Interventions: Drug: Placebo
- Multiple Dose RO7105705 IV (Experimental): Healthy participants or participants with Alzheimer's disease will receive multiple doses of RO7105705 IV QW, a total of 4 doses.
  Interventions: Drug: RO7105705
- Single Dose RO7105705 SC (Experimental): Healthy participants will receive a single dose of RO7105705 SC on Day 1.
  Interventions: Drug: RO7105705
- Single dose Placebo IV (Placebo Comparator): Healthy participants will receive a single dose of placebo IV on Day 1.
  Interventions: Drug: Placebo
- Single dose RO7105705 IV (Experimental): Healthy participants will receive a single dose of RO7105705 IV on Day 1.
  Interventions: Drug: RO7105705

INTERVENTIONS:
Drug: Placebo — Participants will receive single or multiple doses of RO7105705 matching placebo IV.
  Arms: Multiple Dose Placebo IV; Single dose Placebo IV
Drug: RO7105705 — Participants will receive single or multiple doses of RO7105705 IV or SC.
  Arms: Multiple Dose RO7105705 IV; Single Dose RO7105705 SC; Single dose RO7105705 IV

SUMMARY:
This is a Phase I, randomized, placebo-controlled, double-blind study to evaluate the safety, tolerability, pharmacokinetics, and preliminary activity of RO7105705 in two participant populations: healthy participants and participants with mild-to-moderate Alzheimer's disease. This study is a single dose, dose-escalation, and multiple dose study comprising approximately six single dose cohorts in healthy participants administered RO7105705, either intravenously (IV) or subcutaneously (SC), and comprising one or more multiple dose cohorts in healthy participants administered RO7105705 IV every week (QW), a total of 4 doses, and one or more multiple dose cohorts in participants with Alzheimer's disease administered RO7105705 IV QW, a total of 4 doses.

ELIGIBILITY:
Inclusion Criteria:

All participants

* Total body weight between 45 and 120 kilogram (kg), inclusive
* Agreement not to donate blood or blood products for transfusion for the duration of the study and for 1 year after final dose of study drug
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), laboratory tests, and vital signs
* Clinical laboratory evaluations (including chemistry panel fasted [fasted at least 8 hours], complete blood count (CBC), and urine analysis) within the reference range for the test laboratory, unless deemed not clinically significant by the investigator
* Negative test for selected drugs of abuse at screening and at check-in
* Agreement to use highly effective contraception measures

Healthy Participants

* Ages 18-80 years inclusive
* No history of symptomatic cognitive decline and no concern about clinically significant cognitive impairment by the participant or by the investigator

Participants who enroll into a cohort that requires lumbar puncture

* No contraindication to lumbar dural puncture, including coagulopathy, concomitant anticoagulation, thrombocytopenia, prior lumbar spinal surgery, or other factor that precludes safe lumbar puncture in the opinion of the investigator

Participants with Alzheimer's disease

* Ages 50-80 years, inclusive
* The participant should be capable of completing assessments either alone or with the help of the caregiver
* Availability of a person (caregiver) who, in the investigator's judgment, has frequent and sufficient contact with the participant and is able to provide accurate information regarding the participant's cognitive and functional abilities, agrees to provide information at clinic visits, which require partner input for scale completion, and signs the necessary consent form
* Adequate visual and auditory acuity, in the investigator's judgment, sufficient to perform the neuropsychological testing
* Clinical diagnosis of probable Alzheimer's disease dementia based on National Institute on Aging-Alzheimer's Association criteria
* Screening mini-mental state examination (MMSE) score of 16-28 points, inclusive
* Screening Clinical Dementia Rating-Global Score (CDR-GS) of 0.5, 1.0, or 2.0
* Positive florbetapir amyloid positron emission tomography (PET) scan by qualitative read
* If already taking cholinesterase inhibitor and/or memantine therapy for Alzheimer's disease, on a stable dose for at least 4 weeks prior to screening. There should be no intent to, discontinue, or alter the dose of any Alzheimer's disease therapy for the duration of the study

Exclusion Criteria:

Any participants

* Pregnant or lactating, or intending to become pregnant within 16 weeks after last dose of study drug
* Participation in a clinical trial within 30 days before randomization; use of any experimental oral therapy within 30 days or 5 half-lives prior to Day 1, whichever is greater; or use of any biologic therapy within 12 weeks or 5 half-lives prior to Day 1, whichever is greater
* Any non-experimental vaccine within 2 weeks of randomization, until 2 weeks after the last dose
* Surgery or hospitalization during the 4 weeks prior to screening
* Planned procedure or surgery during the study
* Blood transfusion within 8 weeks prior to screening
* Donation or loss of blood (excluding the volume of blood that will be drawn during screening procedures) as follows: 50-499 milliliters (mL) of blood within 30 days or greater than (>) 499 mL of blood within 56 days prior to study drug administration
* Poor peripheral venous access
* Positive for hepatitis C virus (HCV) antibody, hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody
* Illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment
* Administration of any herbal or nutritional supplements (with the exception of standard vitamins and calcium supplements) within 7 days prior to study dose
* Past history of seizures, prior traumatic brain injury, schizophrenia, schizoaffective disorder, or bipolar disorder
* At risk of suicide in the opinion of the investigator
* Serious infection requiring oral and IV antibiotics within 30 days prior to screening
* Any serious medical condition or abnormality in clinical laboratory tests; systemically, clinically immunocompromised because of continuing effects of immune-suppressing medication

Participants with Alzheimer's disease

* History or presence of clinically evident vascular disease potentially affecting the brain
* History or presence of stroke within the previous 2 years or documented history of transient ischemic attack within the previous 12 months
* History or presence of intracranial tumor that is clinically relevant in the opinion of the investigator
* Presence of infections that affect brain function or history of infections that resulted in neurologic sequelae
* History or presence of central nervous system (CNS) or systemic autoimmune disorders potentially causing progressive neurologic disease with associated cognitive deficits
* History or presence of a neurologic disease other than Alzheimer's disease that may affect cognition
* Magnetic resonance imaging (MRI) evidence of 1) more than two lacunar infarcts, 2) any territorial infarct less than (>) 1 centimeters (cm), or 3) significant fluid attenuated inversion recovery (FLAIR) hyperintense lesions in the cerebral white matter that may, in the investigator's opinion, contribute to cognitive dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-06-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Screening up to Day 134
Number of Participants with Dose Limiting Adverse Events (DLAEs) | Day 1 up to Day 36
Change from Baseline in Suicidal Ideation and Behavior Using the Columbia Suicide Severity Rating Scale (C-SSRS) Score | Baseline, up to approximately 134 days

SECONDARY OUTCOMES:
Change From Baseline to Week 19 in Global Function as Assessed Using the Clinical Dementia Rating (CDR) Global Score in Alzheimer's Disease Participants | Baseline, Week 19
Percentage of Participants with Anti-Therapeutic Antibodies (ATAs) | Baseline, Days 29, 57, 113
Serum Concentration of RO7105705 - Single Dose Cohorts: IV Administration | Pre-dose, end of infusion (60-90 minutes), Hour 4, 8, 12 on Day 1, Days 2, 3, 8, 15, 29, 43, 57, 85, 113
Serum Concentration of RO7105705 - Single Dose Cohorts: SC Administration | Pre-dose, Hour 4, 8, 12 on Day 1, Days 2, 3, 4, 6, 8, 15, 29, 43, 57, 85, 113
Serum Concentration of RO7105705 - Multiple Dose Cohorts: IV Administration | Pre-dose, end of infusion (60-90 minutes), Hour 4, 8, 12 on Days 1, 8 15, 22, Days 2, 3, 23, 29, 36, 50, 64, 78, 106, 134
Change From Baseline to Week 19 in Cognitive Function as Assessed Using the Mini-Mental State Examination (MMSE) in Alzheimer's Disease Participants | Baseline, Week 19

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- New Orleans Center for Clinical Research, Knoxville, Tennessee, United States

REFERENCES:
- [Derived] Schauer SP, Toth B, Lee J, Honigberg LA, Ramakrishnan V, Jiang J, Kollmorgen G, Bayfield A, Wild N, Hoffman J, Ceniceros R, Dolton M, Bohorquez SMS, Hoogenraad CC, Wildsmith KR, Teng E, Monteiro C, Anania V, Yeh FL. Pharmacodynamic effects of semorinemab on plasma and CSF biomarkers of Alzheimer's disease pathophysiology. Alzheimers Dement. 2024 Dec;20(12):8855-8866. doi: 10.1002/alz.14346. Epub 2024 Nov 8. PMID 39513754